CLINICAL TRIAL: NCT01765764
Title: Bimatoprost for the Treatment of Eyebrow Hypotrichosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-043
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Eyebrow Hypotrichosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bimatoprost Solution BID (Experimental): Bimatoprost solution twice a day (BID) in the morning and in the evening applied to each eyebrow for 7 months.
  Interventions: Drug: bimatoprost solution
- Bimatoprost Solution QD (Experimental): Vehicle to bimatoprost solution in the morning and bimatoprost solution once a day (QD) in the evening applied to each eyebrow for 7 months.
  Interventions: Drug: bimatoprost solution; Drug: Vehicle to bimatoprost solution
- Vehicle to Bimatoprost Solution BID (Placebo Comparator): Vehicle to bimatoprost twice a day (BID) in the morning and the evening applied to each eyebrow for 7 months.
  Interventions: Drug: Vehicle to bimatoprost solution

INTERVENTIONS:
Drug: bimatoprost solution — Bimatoprost solution once a day or twice a day applied to each eyebrow for 7 months.
  Arms: Bimatoprost Solution BID; Bimatoprost Solution QD
Drug: Vehicle to bimatoprost solution — Vehicle to bimatoprost solution once or twice a day applied to each eyebrow for 7 months.
  Arms: Bimatoprost Solution QD; Vehicle to Bimatoprost Solution BID

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost solution compared with vehicle in the treatment of eyebrow hypotrichosis (inadequate eyebrows).

ELIGIBILITY:
Inclusion Criteria:

-Adult participants with eyebrow hypotrichosis (inadequate eyebrow growth).

Exclusion Criteria:

* Patients with disease, infection, or abnormality of the eyebrow area
* Patients with permanent eyebrow loss due to over-grooming

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Houston, Texas, United States
- Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Carruthers J, Beer K, Carruthers A, Coleman WP 3rd, Draelos ZD, Jones D, Goldman MP, Pucci ML, VanDenburgh A, Weng E, Whitcup SM. Bimatoprost 0.03% for the Treatment of Eyebrow Hypotrichosis. Dermatol Surg. 2016 May;42(5):608-17. doi: 10.1097/DSS.0000000000000755. PMID 27124878

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Started | 118 | 118 | 121
Completed | 115 | 109 | 115
Not Completed | 3 | 9 | 6
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Personal Reasons | 1 | 2 | 1
Not completed — Other Miscellaneous Reasons | 1 | 2 | 2
Period: Post-treatment Period
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Started | 114 (1 participant did not enter the Post-treatment Period. [Personal Reasons]) | 107 (2 participants did not enter the Post-treatment Period [2 Lost-to-Follow-up (LFU)]) | 112 (3 participants did not enter the Post-treatment Period [1 Personal Reasons,2 LFU].)
Completed | 114 | 107 | 112
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID | Total
Number analyzed (Participants) | 118 | 118 | 121 | 357
Age, Customized [Number; unit: Participants]
  18 to <45 years | 18 | 19 | 22 | 59
  ≥45 years | 100 | 99 | 99 | 298
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 112 | 112 | 338
  Male | 4 | 6 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-Grade Increase (Improvement) in the 4-Point Global Eyebrow Assessment (GEBA) Scale
Description: The physician evaluated eyebrow fullness using the 4-point GEBA Scale where: 1=very sparse, 2=sparse, 3=full and 4=very full. The percentage of participants with at least a 1-grade increase from Baseline is reported.
Time Frame: Baseline, Month 7
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Number analyzed (Participants) | 118 | 118 | 121
percentage of participants | 83.9 | 77.1 | 43.0

2. Secondary Outcome: Change From Baseline in Eyebrow Fullness as Measured Using Digital Monitoring System Image Analysis (DMSIA)
Description: Photographs were taken of the eyebrows. Eyebrow fullness was measured by DMSIA for both eyes and averaged. Eyebrow fullness was reported in millimeters squared (mm^2). A positive change from Baseline indicated fuller eyebrows (improvement).
Time Frame: Baseline, Month 7
Population: Participants from the Intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Number analyzed (Participants) | 117 | 117 | 118
mm^2
  Baseline | 101.08 (47.252) | 97.80 (41.525) | 98.17 (49.657)
  Change from Baseline at Month 7 | 34.51 (35.940) | 30.96 (33.638) | 6.42 (26.870)

3. Secondary Outcome: Change From Baseline in Eyebrow Darkness as Measured Using DMSIA
Description: Photographs were taken of the eyebrows. Eyebrow darkness (intensity) was measured by DMSIA for both eyes and averaged. Eyebrow darkness was reported in intensity units. A negative change from Baseline indicated darker eyebrows (improvement).
Time Frame: Baseline, Month 7
Population: Participants from the Intent-to-treat population, all randomized participants, with data available for analysis.
Measure: Mean (Standard Deviation); unit: intensity units
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Number analyzed (Participants) | 116 | 116 | 117
intensity units
  Baseline | 53.90 (6.314) | 53.59 (7.688) | 52.87 (6.985)
  Change from Baseline at Month 7 | -4.53 (3.294) | -3.76 (3.212) | 0.11 (1.837)

4. Secondary Outcome: Percentage of Participants With 'Very Satisfied' or 'Mostly Satisfied' in Eyebrow Satisfaction Scale (ESS) Item #6
Description: ESS Item #6 measured the participant's satisfaction with eyebrow treatment: "Overall, how satisfied are you with the way the eyebrow treatment makes your eyebrows look right now?" using a 5-point scale where: 1=very satisfied, 2=mostly satisfied, 3=neither dissatisfied nor satisfied, 4=mostly dissatisfied and 5=very dissatisfied. The percentage of participants 'very satisfied' or 'mostly satisfied' is reported.
Time Frame: Month 7
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Number analyzed (Participants) | 118 | 118 | 121
percentage of participants | 70.3 | 52.5 | 36.4

ADVERSE EVENTS:
Arm/Group | Bimatoprost Solution BID | Bimatoprost Solution QD | Vehicle to Bimatoprost Solution BID
Serious Adverse Events (participants affected / at risk) | 2/118 | 0/118 | 5/121
Other Adverse Events (participants affected / at risk) | 6/118 | 5/118 | 7/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Solution BID (N=118) | Bimatoprost Solution QD (N=118) | Vehicle to Bimatoprost Solution BID (N=121)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Solution BID (N=118) | Bimatoprost Solution QD (N=118) | Vehicle to Bimatoprost Solution BID (N=121)
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.